CLINICAL TRIAL: NCT00360074
Title: A Randomised, Controlled, Crossover Study: Treatment With Thyroxin Compared to Thyroxin + Triiodothyronin in Patients With Secondary Hypothyroidism
Brief Title: Phase 4 Study in Secondary Hypothyroidism: Body Weight Adapted Thyroxin Treatment and Triiodothyronine Supplementation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital Freiburg (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: FH 326/03
Record Dates: First submitted 2006-08-02; First posted 2006-08-03 (Estimated); Last update posted 2008-06-09 (Estimated); Status verified 2008-06

CONDITIONS: Secondary Hypothyroidism; Hypopituitarism; Hyperlipidemias
Keywords: secondary hypothyroidism; body weight adjusted thyroxin dose; triiodothyronine supplementation
MeSH Terms: conditions — Hypothyroidism; Hypopituitarism; Hyperlipidemias | interventions — Thyroxine; Triiodothyronine

INTERVENTIONS:
Drug: Thyroxin, Triiodothyronine

SUMMARY:
The purpose of this study is to determine whether a body weight adjusted dose of thyroxin is superior to treatment guided by laboratory results of thyroxin hormones in patients with central hypothyroidism. Moreover beneficial effects of triiodthyronine supplementation are investigated.

DETAILED DESCRIPTION:
Backround: A normal thyroid function is critical for metabolism, well-being and cognitive function. It is now well accepted that primary subclinical hypothyroidism, characterized by normal circulating thyroid hormones (fT3 and fT4) and elevated TSH, should be treated to improve reduced quality of life and abnormalities of lipid metabolism. In central hypothyroidism (CH) the dose of replacement therapy aims to achieve normal thyroxin (T4) concentrations as defined by appropriate reference populations. Adequate thyroxin treatment is especially challenging, as T4 cannot be titrated according to endogenous TSH levels because of the impaired hypothalamic-pituitary unit. The majority of untreated CH patients show normal (40 %) or elevated TSH levels (35 %) while only a minority has reduced concentrations (25 %) {Faglia, 1979 #1}. These findings are explained by the lack of pulsatile secretion and nocturnal TSH surge, which has been attributed to impaired thyrotroph function in CH patients {Caron, 1986 #2}. Moreover, impaired biological activity of TSH itself due to reduced glycosylation has been described in secondary hypothyroidism.

In a cross sectional study performed in patients with central hypothyroidism, we found elevated cholesterol levels and increased ankle reflex time suggesting subtle hypothyroidism, though fT3 and fT4 serum concentrations were within the normal range. The average dose of thyroxin (T4) applied in these patients with central hypothyroidism was 1.1 µg/kg bw, which is below the average dose recommended in primary hypothyroidism (1.6 µg/kg bw). We hypothesized that these results might indicate suboptimal T4 replacement therapy, not detectable by current laboratory testing.

Hypothesis: To investigate the effects of a body weight adjusted T4 or T3T4 dose on metabolism, well-being and cognitive function.

Study design: Placebo controlled trial in patients with central hypothyroidism following a double blind cross-over design.

Intervention: Three different treatment regimes (5 weeks each) were compared: "CON-T4", empirically chosen, current dose of T4 (1 ± 0.05 μg/kg body weight (bw); "OPT-T4", optimized T4 treatment (1.6 μg/kg bw T4); "T3T4", combination of triiodothyronine (T3, 0.16) and T4 (1.44 μg/kg bw). Biochemical parameters, ankle reflex time and neurocognitive functions were assessed.

ELIGIBILITY:
Inclusion Criteria:

* hypopituitarism of at least 3 axes (TSH plus gonadotropin, somatotropin, corticotropin or ADH deficiency)
* termination of surgical or radiation treatment of pituitary tumors at least six month before study entry
* BMI of 20 - 39.9 kg/m2
* non-smoking status.

Exclusion Criteria:

* history of cardiovascular or pulmonary diseases
* current thyroxin dosage > 1.6 µg/kg bw
* pregnancy
* epilepsy
* cerebrovascular diseases
* nodular goiter

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25
Dates: Start 2004-02; Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
well-being | 3 weeks of treatment
cognitive function | 3 weeks of treatment

SECONDARY OUTCOMES:
lipid metabolism | 3 weeks of treatment
muscle function / ankle reflex time | 3 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Prof Dr Martin Reincke, MD, Principal Investigator — former Medical Professor of University Hospital Freiburg
Locations (1):
- University Hospital Freiburg, Department of Medicine, Freiburg im Breisgau, Baden-Wurttemberg, Germany

REFERENCES:
- [Result] Slawik M, Klawitter B, Meiser E, Schories M, Zwermann O, Borm K, Peper M, Lubrich B, Hug MJ, Nauck M, Olschewski M, Beuschlein F, Reincke M. Thyroid hormone replacement for central hypothyroidism: a randomized controlled trial comparing two doses of thyroxine (T4) with a combination of T4 and triiodothyronine. J Clin Endocrinol Metab. 2007 Nov;92(11):4115-22. doi: 10.1210/jc.2007-0297. Epub 2007 Aug 21. PMID 17711927